CLINICAL TRIAL: NCT00351871
Title: Influence of Marker of Insulin Resistance Upon HCV Treatment Responses to PEG Intron and Rebetol Therapy
Brief Title: Influence of Marker of Insulin Resistance Upon Hepatitis C Virus (HCV) Treatment Responses to PEG Intron and Rebetol Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03851
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

INTERVENTIONS:
Drug: PEG-Intron Plus REBETOL

SUMMARY:
The objective of this study is to better understand the influence of insulin resistance upon treatment response in hepatitis C virus treated with PEG Intron and Rebetol.

DETAILED DESCRIPTION:
The relationship between HCV and IR is an evolving one. This study will allow a more formal evaluation of this relationship. Four hundred patients will be treated using weight based Peg Intron and Rebetol. Clinical and biochemical data related to IR will be collected to determine if any such factors can predict who will have a sustained virological response. To evaluate patients for insulin resistance, the HOMA score (the product of the fasting insulin level and blood glucose level), waist circumference, and body mass index will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of chronic hepatitis C infection (viremia) by RT-PCR superquantitative
* HCV Genotype 1
* Liver biopsy within 36 months of enrollment consistent with chronic hepatitis
* Compensated liver disease with laboratory parameters at entry visit as follows:

  * Hemoglobin values of > 12 gm/dL
  * WBC > 2,500/mm3
  * Neutrophil count > 1,000/mm3
  * Platelets > 100,000/mm3
  * Prothrombin time < 2 seconds prolonged compared to control, or equivalent INR ratio
* Bilirubin within 20% of the upper limit of normal unless non-hepatitis related factors exists such as Gilbert's syndrome.
* Albumin > 3.0 g/dL
* Serum creatinine < 1.4 mg/dL
* Normal thyroid stimulating hormone (TSH) or thyroid disease clinically controlled
* Antinuclear antibodies (ANA)< 1:160
* FBS < 126 mg/dl
* No significant co-existing psychiatric disease
* Free from substance abuse for past 2 years

Exclusion Criteria:

* Previous treatment for HCV.
* Evidence of being HIV positive.
* Hypersensitivity to alpha interferon, Peg Intron or Rebetol.
* Any other causes for chronic liver disease other than chronic hepatitis C besides obesity.
* Hemoglobinopathies (e.g., Thalassemia) or any other cause of hemolytic anemia.
* Evidence of advanced liver disease such as a history of or presence of ascites, bleeding varices, or hepatic encephalopathy.
* Preexisting medical condition that could interfere with the patient's participation in the protocol including: CNS trauma or active seizure disorders requiring medication; diabetes mellitus; serious pulmonary disease; immunologically mediated diseases; gout attack within 12 months; or any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.
* Patients with evidence of ischemia on stress testing, an arrhythmia, cardiac failure, coronary surgery, uncontrolled hypertension, angina or a myocardial infarction within 12 months.
* Patients with a history of organ transplantation will be excluded.
* Patients taking insulin sensitizing drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Difference in treatment response rates between those with insulin resistance those without.

SECONDARY OUTCOMES:
Which marker of Insulin Resistance (i.e. the HOMA score, Waste Circumference or BMI) is the best measure for risk of hypo responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: William M. Cassidy, M.D., Principal Investigator — Louisiana State University Health Sciences Center